CLINICAL TRIAL: NCT01694420
Title: Treatment of Acute HIV Infection With the Elvitegravir, Cobicistat, Emtricitabine, and Tenofovir Disoproxil Fumarate, A Pilot Study of Response to Therapy and HIV Pathogenesis
Brief Title: Treatment of Acute HIV Infection With Quad Fixed-dose Combination (FDC) Tablet
Acronym: PHI04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00035447; IN-US-236-0124 (Other Grant/Funding Number: Funder)
Record Dates: First submitted 2012-09-21; First posted 2012-09-27 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: HIV
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quad FDC (Experimental): FDC elvitegravir + cobicistat + tenofovir + emtricitabine STR once daily for 48 weeks
  Interventions: Drug: (FDC) ELV/COBI/FTC/TDF

INTERVENTIONS:
Drug: (FDC) ELV/COBI/FTC/TDF — Antiretroviral treatment
  Other Names: STRIBILD

SUMMARY:
This is a multicenter, single arm, 48-week open-label study of FDC ELV/COBI/FTC/TDF [Stribild] in acute HIV infection. Study sites will be members of the Duke-UNC Acute HIV Infection Study Consortium. Participants will be enrolled for 96 weeks. Clinical care and study drug (ELV/COBI/FTC/TDF) will be provided for the first 48 weeks. After week 48, clinical care but not study drug will be provided through week 96. A study participant suppressed at week 48 can continue on FDC ELV/COBI/FTC/TDF.

The primary hypothesis is that once daily fixed-dose combination elvitegravir (ELV), cobicistat (COBI), emtricitabine (FTC), and tenofovir disoproxil fumarate (TDF) will rapidly reduce viral replication to <50 copies RNA/ml in participants with acute HIV infection. The secondary hypotheses to be considered are 1) virologic response rates as measured by plasma HIV RNA levels will be non-inferior or superior to a historical group of participants from the PHI cohort treated with EFV/FTC/TDF, 2) compared to historical controls treated with EFV/FTC/TDF, plasma HIV RNA will decrease more rapidly in PHI participants treated with ELV/COBI/FTC/TDF, 3) compared to historical controls treated with EFV/FTC/TDF, immune activation as measured by the proportion CD4+ and CD8+ cells expressing HLA-DR and CD38+ will decrease more rapidly in PHI participants treated with ELV/COBI/FTC/TDF, 4)in a subset of participants samples will be obtained from compartments such as the gastrointestinal tract, and lymphoid tissues to assess changes over time in parameters such as HIV-1 RNA, immunologic responses to HIV, and tissue and anatomic reservoirs. We hypothesize that treatment with the ELV/COBI/FTC/TDF will demonstrate improved viral clearance in these compartments as compared to historical controls treated with EFV/FTC/TDF. 5) in a subset of participants who remain suppressed on therapy, resting CD4 cells with replication-competent HIV-1 (latent reservoir) will be quantitated and compared to similar measurements in PHI participants treated with EFV/FTC/TDF. In addition, we will compare these results to those measured in HIV-1 infected participants treated and 6) ELV/COBI/FTC/TDF will be well tolerated, and the proportion of participants who require treatment modification will be less than that observed in participants treated with EFV/FTC/TDF.

DETAILED DESCRIPTION:
None desired

ELIGIBILITY:
Acute HIV infection is defined as:

1. A positive 4th generation HIV Ag/Ab Combination Assay and HIV RNA (NAAT or viral load) and one of the following within 30 days of study entry:

   * a negative HIV rapid test
   * negative/indeterminate Western Blot

   OR
2. A negative or indeterminate HIV antibody, antigen, or nucleic acid amplification test (NAAT) and any one of the following within 30 days of study entry:

   * A detectable HIV nucleic acid in blood confirmed by a second NAAT
   * Positive p24 antigen
   * A positive HIV antibody test according to standard criteria obtained within 45 days after an initial negative or indeterminate HIV antibody, antigen, or nucleic acid amplification.

Inclusion Criteria:

1. Acute HIV Infection (as defined above) within 30 days of study entry.
2. Age >18 years.
3. ART-naive (<14 days of previous antiretroviral treatment. Exceptions are: Post-exposure prophylaxis (PEP) if participant was documented as HIV-negative at least 3 months after completion of PEP.
4. Lab values within 30 days prior to study entry:

   1. Absolute neutrophil count >500/mm3
   2. Hemoglobin > 8.5 g/dL for men and > 8.0 g/dL for women
   3. Platelet count >50,000/mm3
   4. AST (SGOT)> .2.5 x ULN
   5. ALT (SGPT)> .2.5 x ULN
   6. Total bilirubin <2.5 x ULN
   7. Calculated creatinine clearance (Cockcroft-Gault formula) > 70mL/min:
5. For women of reproductive potential, a negative pregnancy test within 72 hours prior to initiating antiretroviral study medications. Reproductive potential is defined as females who have reached menarche and have not been post-menopausal for at least 24 consecutive months, or have not undergone surgical sterilization.
6. Female study participants must use a reliable form of barrier contraception, such as a condom, even if they also use other methods of birth control. All participants must continue to use contraception for 12 weeks after stopping study medications. Acceptable methods of barrier contraception include: condoms (male or female), diaphragm, or cervical cap. These can be used alone or in tandem with hormonal or IUD method.
7. Ability and willingness of participant to give written informed consent.

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Women with a positive pregnancy test prior to study drug administration.
3. Men who have sex with women, and women of reproductive potential unwilling or unable to use an acceptable, reliable barrier method of contraception for the entire study period and 12 weeks afterwards.
4. Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days of study entry (Prednisone 10 mg QD or less is permitted.
5. Known allergy/sensitivity to study drugs
6. Difficulty swallowing pills
7. Inability to communicate effectively with study personnel
8. Incarceration; prisoner recruitment and participation are not permitted
9. Active drug or alcohol use that, in the opinion of the site investigator, would interfere with participation in the study
10. Any active psychiatric illness that, in the opinion of the investigator, could confound the analysis of the neurological examination or neuropsychological test results
11. Active brain infection (except for HIV-1), brain neoplasm, space-occupying brain lesion requiring acute or chronic therapy
12. Serious illness requiring systemic treatment and/or hospitalization until patient either completes therapy or is clinically stable on therapy for at least 7 days prior to study entry
13. Known cardiac conduction disease
14. Prior treatment with any other experimental drug within 30 days of initiating study treatment
15. Unable to discontinue any current medications that are excluded during study treatment
16. Life expectancy less than twelve months
17. Acute Viral Hepatitis, including, but not limited to, Hepatitis A, B, or C
18. Chronic Hepatitis B Infection documented by a detectable serum Hepatitis B surface antigen (HBsAg) or plasma HBV DNA
19. Calculated creatinine clearance (Cockcroft-Gault formula) <70mL/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2016-04 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehri McKellar, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - UNC at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Gay CL, Mayo AJ, Mfalila CK, Chu H, Barry AC, Kuruc JD, McGee KS, Kerkau M, Sebastian J, Fiscus SA, Margolis DM, Hicks CB, Ferrari G, Eron JJ; Duke-UNC Acute HIV Infection Consortium. Efficacy of NNRTI-based antiretroviral therapy initiated during acute HIV infection. AIDS. 2011 Apr 24;25(7):941-9. doi: 10.1097/QAD.0b013e3283463c07. PMID 21487250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this study are recruited from AHI participants referred to our ID clinics. Referrals are generated from the NC STAT Program and from clinical diagnoses made by both internal and external health care clinics.
Period: Overall Study
Arm/Group | Quad FDC
Started | 33
Completed | 30
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Quad FDC
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Viral Load Measurement of <200 Copies/mL at Week 24
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Quad FDC
Number analyzed (Participants) | 30
participants | 28

2. Primary Outcome: Virologic Efficacy of the Fixed Dose Combination (FDC) ELV/COBI/FTC/TDF Given Once Daily to Participants With Acute HIV Infection as Determined by the Proportion of Treated Participants With HIV-1 RNA to <50 Copies/mL at Week 48
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Quad FDC
Number analyzed (Participants) | 30
participants | 24

3. Secondary Outcome: Immune Activation as Measured by the Proportion of CD4+ and CD8+ Cells Expressing HLA-DR and CD38+
Time Frame: 48 weeks
Population: Data not collected
Arm/Group | Quad FDC
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Virologic Decline in the First 48 Weeks of Treatment Comparing FDC ELV/COBI/FTC/TDF to FDC EFV/FTC/TDF
Time Frame: 48 weeks
Measure: Median (Full Range); unit: days
Arm/Group | Quad FDC
Number analyzed (Participants) | 30
days
  HIV RNA <200 copies/mL | 26 [7 to 132]
  HIV RNA <50 copies/mL | 54 [12 to 251]
Statistical Analysis 1: Comparison: Quad FDC; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Study data compared to data as cited in PubMed ID: 21487250

5. Other Pre Specified Outcome: Number of Participants With Grade 3 or Grade 4 Adverse Events
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Quad FDC
Number analyzed (Participants) | 30
participants
  Grade 3 | 3
  Grade 4 | 0

6. Other Pre Specified Outcome: Number of Participants With Adverse Events Related to Study Drug
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Quad FDC
Number analyzed (Participants) | 30
participants | 22

ADVERSE EVENTS:
Arm/Group | Quad FDC
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 22/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quad FDC (N=33)
Anemia (Blood and lymphatic system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Chest wall injury (Injury, poisoning and procedural complications) | 1
Constipation (Gastrointestinal disorders) | 1
Decreased appetite (General disorders) | 1
Decreased comprehension (Nervous system disorders) | 1
Decreased neutrophils (Blood and lymphatic system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Disseminated itching (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry mouth (General disorders) | 1
Elevated ALT (Hepatobiliary disorders) | 4
Elevated AST (Hepatobiliary disorders) | 5
Elevated BP during leukapheresis (Surgical and medical procedures) | 7
Elevated creatinine (Renal and urinary disorders) | 1
Elevated lipase (Hepatobiliary disorders) | 1
Elevated cholesterol (Endocrine disorders) | 1
Fatigue (General disorders) | 5
Feeling of air stuck in throat (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 7
Hot flashes (General disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Increased appetite (Gastrointestinal disorders) | 1
Alteration in taste (General disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Night sweats (General disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Shigella colitis (Gastrointestinal disorders) | 2
Short term memory loss (Nervous system disorders) | 1
stomach cramping (Gastrointestinal disorders) | 1
thigh weakness (General disorders) | 1
thinning hair (Skin and subcutaneous tissue disorders) | 1
Tingling around lips during leukaphersis (Surgical and medical procedures) | 4
Weight loss (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No